CLINICAL TRIAL: NCT03797833
Title: Spinal Anesthesia for External Cephalic Version in Nulliparous Women, A Controlled Randomized Study
Brief Title: Spinal Anesthesia for External Cephalic Version
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow inclusion rate. Central contact person quit for another job.
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018/634
Record Dates: First submitted 2019-01-07; First posted 2019-01-09 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Breech Presentation; Before Labor
Keywords: breech presentation, external version, spinal anaesthesia
MeSH Terms: conditions — Breech Presentation | interventions — Anesthesia, Spinal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard treatment (No Intervention): ECV according to standard practice.
- Spinal anaesthesia (Active Comparator): ECV after low dose spinal anaesthesia (Bupivacain 2,5 mg plus Sufentanil 5 micrograms (µg)
  Interventions: Procedure: Spinal Anaesthesia

INTERVENTIONS:
Procedure: Spinal Anaesthesia — Spinal anaesthesia with Bupivacain 2.5 mg and Sufentanil 5 µg
  Arms: Spinal anaesthesia

SUMMARY:
This study evaluates the potential benefits of spinal anaesthesia for nulliparous mothers scheduled for external version of babies in breech position.

DETAILED DESCRIPTION:
Fetuses in breech position are almost always delivered by Caesarian section (CS). If the fetus is in breech position by the end of pregnancy, attempts for external cephalic version (ECV) are usually made. The success rate of ECV in nulliparous women is lower than in multiparous women. There are studies showing a higher rate of successful ECV's if the mother received a low dose spinal anaesthesia (SA). Overall maternal satisfaction was higher with SA. These studies, however, did not take parity into account.

The primary aim of this study is to see if SA can increase the rate of successful ECV's in nulliparous women.

The secondary aims are to evaluate if maternal satisfaction increases and if the rate of CS is decreasing using SA during ECV.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant nulliparous women.
* Breech presentation of fetus, eligible for external version.

Exclusion Criteria:

* Unwilling to participate.
* Unable to understand written and oral Swedish in the absence of interpreter.
* Contraindications to spinal anaesthesia.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-01-07 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
External version success rate | 1 hour
  Rate of successful version as assessed by gynaecologist after maximum three attempts.

SECONDARY OUTCOMES:
Overall maternal satisfaction post external version attempt | 1 hour
  Evaluation of overall participant satisfaction using an online assessment questionnaire within an hour from the external version attempts.
Overall maternal satisfaction post partum | 3 months
  Evaluation of overall participant satisfaction using an online assessment questionnaire within 3 months from the external version attempts (within 2 months post partum)
Caesarian section rate | 1 months
  The mode of delivery, assessed from the medical charts after delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Herbst, MD PhD, Principal Investigator — Lund University, IKVL gyn/ob . Skåne University Hospital, Lund Sweden
Locations (2):
- Sweden (2):
  - Skåne University Hospital, Lund
  - Skåne University Hospital, Malmo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Khaw KS, Lee SW, Ngan Kee WD, Law LW, Lau TK, Ng FF, Leung TY. Randomized trial of anaesthetic interventions in external cephalic version for breech presentation. Br J Anaesth. 2015 Jun;114(6):944-50. doi: 10.1093/bja/aev107. Epub 2015 May 10. PMID 25962611
- [Background] Magro-Malosso ER, Saccone G, Di Tommaso M, Mele M, Berghella V. Neuraxial analgesia to increase the success rate of external cephalic version: a systematic review and meta-analysis of randomized controlled trials. Am J Obstet Gynecol. 2016 Sep;215(3):276-86. doi: 10.1016/j.ajog.2016.04.036. Epub 2016 Apr 27. PMID 27131581
- [Background] Cluver C, Gyte GM, Sinclair M, Dowswell T, Hofmeyr GJ. Interventions for helping to turn term breech babies to head first presentation when using external cephalic version. Cochrane Database Syst Rev. 2015 Feb 9;2015(2):CD000184. doi: 10.1002/14651858.CD000184.pub4. PMID 25674710
- [Background] Chalifoux LA, Bauchat JR, Higgins N, Toledo P, Peralta FM, Farrer J, Gerber SE, McCarthy RJ, Sullivan JT. Effect of Intrathecal Bupivacaine Dose on the Success of External Cephalic Version for Breech Presentation: A Prospective, Randomized, Blinded Clinical Trial. Anesthesiology. 2017 Oct;127(4):625-632. doi: 10.1097/ALN.0000000000001796. PMID 28723831